CLINICAL TRIAL: NCT02586675
Title: The TEEL Study: A Phase I Trial of Tamoxifen With Ribociclib (LEE011) in Adult Patients With Advanced ER+ (HER2 Negative) Breast Cancer
Brief Title: TEEL Study- Phase 1 Tamoxifen and Ribociclib (LEE011) in Advanced ER+ (HER2 Negative) Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-18332
Record Dates: First submitted 2015-10-23; First posted 2015-10-26 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Breast Cancer; Breast Cancer - Female; Breast Cancer - Male
Keywords: ER+ breast cancer; PR+ breast cancer; hormone receptor positive; HER2- breast cancer; HER2 negative; locally advanced; metastatic
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male; Neoplasm Metastasis | interventions — Tamoxifen; ribociclib; Cyclin-Dependent Kinases; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tamoxifen and Ribociclib with Goserelin (Experimental): Phase I dose escalation followed by Phase Ib dose expansion. Tamoxifen and Ribociclib, with Goserelin added for premenopausal or peri-menopausal participants. Ribociclib: Capsules/Tablets for oral use 400 mg OR 600 mg Days 1-21 of each 28 day cycle or daily. Tamoxifen: Tablets for oral use 20 mg daily (all days of every cycle without interruption). Goserelin: Subcutaneous injection 3.6 mg Day 1 of each 28 day cycle.
  Interventions: Drug: Tamoxifen; Drug: Ribociclib; Drug: Goserelin

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen will be taken orally once daily on a continuous daily schedule (e.g., days 1-28 of each 28 day cycle).
Drug: Ribociclib — Ribociclib (LEE011) will be taken orally once daily on days 1-21 of each 28 day cycle. Days 22-28 will be a "rest" period from dosing with Ribociclib. In the continuous cohort, 400 mg ribociclib will be given daily (QD).
  Other Names: LEE011; Cyclin-Dependent Kinase (CDK) Inhibitor
Drug: Goserelin — Goserelin will be given as an injectable subcutaneous implant on day 1 of every 28 day cycle. This will be given in pre-menopausal and peri-menopausal women.
  Other Names: Zoladex; Goserelin acetate

SUMMARY:
The purpose of this study is to find out if the investigational drug Ribociclib (LEE011), when taken with standard treatment (Tamoxifen +/- Goserelin) is safe and has beneficial effects in pre-menopausal and post-menopausal women and men who have a type of breast cancer known as hormone receptor positive/HER2- breast cancer.

DETAILED DESCRIPTION:
Phase I Dose Escalation:

The phase I portion of the study is a dose escalation to confirm the safety of the combination and to determine the Maximum Tolerated Dose (MTD) and the Recommended Phase II Dose (RP2D) for ribociclib with Tamoxifen.

Phase I will be conducted in all participants with Hormone Receptor Positive (HR+)/Human Epidermal growth factor Receptor 2 Negative (HER2-) locally advanced or metastatic breast cancer with any prior endocrine therapy and up to three prior cytotoxic chemotherapy regimens administered in the metastatic or locally advanced setting.

Phase Ib Dose Expansion:

Phase I trials are increasingly including dose-expansion cohorts (Ib) after the maximum-tolerated dose has been reached to better characterize the toxicity profile and identify early signs of efficacy within this specific disease population. The investigators' goal is to assess the anti-tumor activity Ribociclib + Tamoxifen and to further evaluate their safety in adult patients with HR+/HER2- locally advanced or metastatic breast cancer. Patients in the phase 1b expansion will have the same exclusion and inclusion criteria except that they will only be allowed to have up to two lines of cytotoxic chemotherapy in the metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

* Histologically and/or cytologically confirmed diagnosis of Estrogen Receptor-Positive (ER+) and/or Progesterone Receptor-Positive (PR+) breast cancer by local laboratory.
* Human Epidermal growth factor Receptor 2 Negative (HER2-) breast cancer defined as a negative in situ hybridization test or an Immunohistochemistry (IHC) status of 0, 1+ or 2+. If IHC is 2+, a negative In Situ Hybridization (Fluorescence [FISH], Chromogenic [CISH], or Silver [SISH]) test is required by local laboratory testing.
* Participants are allowed (but not required) to have up to two lines of prior chemotherapy regimens in the metastatic setting for the dose expansion phase. For the dose escalation cohort, up to three previous lines of chemotherapy in the metastatic setting is acceptable.
* Measurable disease, i.e., at least one measurable lesion as per Response Evaluation Criteria in Solid Tumors (RECIST)1.1 criteria only *for expansion cohorts.
* For *escalation cohorts, bone only disease is allowed. For expansion cohorts, there must be measurable disease as stated above.
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 or 1.
* Written informed consent must be obtained prior to any screening procedures and according to local guidelines.
* Adequate bone marrow and organ function.
* Must be able to swallow ribociclib and Tamoxifen capsules/tablets.
* Pre-Menopausal Women Eligibility: 1) Pre-menopausal women who received adjuvant Aromatase Inhibitor and Ovarian Suppression (AI + OS) in the adjuvant setting and completed at least 12 months of hormonal therapy. 2) Pre-menopausal women with de novo metastatic disease are eligible if they have had no prior endocrine therapy. 3) Pre-menopausal women who have not received Tamoxifen in the metastatic setting, but have received up to two lines of chemotherapy.
* Post-Menopausal Women and Men Eligibility: 1) Post-menopausal women or men who have progressed on first-line or second line therapy with an aromatase inhibitor in the metastatic setting. 2) Post-menopausal women or men who have recurred while on or after completion of adjuvant treatment with aromatase inhibitors (they have completed at least one year of AI in the adjuvant setting before progression on AI). 3) Post-menopausal women or men who are not considered candidates for treatment with an aromatase inhibitory by their oncologist, patients not willing to go on AI, or patients who were intolerant to AI.
* Post-menopausal women or men are allowed (but not required) to have up to two lines of prior chemotherapy regimens in the metastatic setting for the dose expansion phase . For the dose escalation cohort, up to three previous lines of chemotherapy in the metastatic setting is acceptable.

Exclusion Criteria:

* Potential participants with inflammatory breast cancer.
* Prior CDK 4/6 inhibitor exposure.
* Have received Tamoxifen in the metastatic setting (for more than 30 days) or has progressed while on Tamoxifen in the adjuvant setting.
* Known hypersensitivity to ribociclib or excipients of tamoxifen.
* A concurrent malignancy or malignancy within 3 years of starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
* Central nervous system (CNS) involvement unless specific criteria are met.
* Impairment of Gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Known history of HIV infection (testing not mandatory).
* Any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Clinically significant, uncontrolled heart disease and/or a recent events as specified in the study protocol
* Currently receiving any of the following medications and cannot be discontinued 7 days prior to starting study drug: a. Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges. b. That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5. c. That have a known risk to prolong the QT interval or induce Torsades de Pointes. d. Herbal preparations/medications, dietary supplements not prescribed by an M.D..
* Currently receiving or has received systemic corticosteroids ≤2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.
* The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
* Currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Participation in a prior investigational study within 30 days prior to enrollment..
* Has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥ 25% of the bone marrow was irradiated.
* Has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
* Has not recovered from all toxicities related to prior anticancer therapies to NCI Common Terminology Criteria for Adverse Events (CTCAE) version 4.03 Grade equal to or less than 1 (Exception to this criterion: patients with any grade of alopecia are allowed to enter the study).
* A Child-Pugh score B or C.
* History of non-compliance to medical regimen or inability to grant consent.
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human Chorionic Gonadotropin (hCG) laboratory test.]
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 12 weeks after study drug discontinuation. There are specific guidelines regarding the various acceptable highly effective contraception methods. Note: The use of oral contraception is not allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-02-23 (Actual); Primary Completion 2017-05-08 (Actual); Study Completion 2021-10-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roohi Ismail-Khan, MD, MSc, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center and Research Institute, Tampa, Florida, United States

REFERENCES:
- See also: Moffitt Cancer Center Clinical Trials website — https://www.moffitt.org/clinical-trials-research/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center March 2016 through September 2016. All participants were enrolled and treated on Cohort 1 (Ribociclib 400 mg PO D1-21; Tamoxifen 20 mg PO QD (1) only.
Period: Overall Study
Arm/Group | Tamoxifen and Ribociclib With Goserelin
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All participants.
Groups:
- Tamoxifen and Ribociclib With Goserelin: Phase I dose escalation followed by Phase Ib dose expansion.
Arm/Group | Tamoxifen and Ribociclib With Goserelin
Number analyzed (Participants) | 7
Age, Continuous [Median (Standard Deviation); unit: years] | 54 (13.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (RP2D)
Description: 400-600 mg of Ribociclib, when taken with Tamoxifen 20 mg. The Phase I portion of the study is a dose escalation to confirm the dose limiting toxicity (DLT) and the RP2D for ribociclib with Tamoxifen. DLT is defined as an adverse event or abnormal laboratory value assessed as having a reasonable possibility related to the study medication, unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first 28 days of treatment (cycle 1) with LEE011 and Tamoxifen. National Cancer Institute Common Terminology Criteria for Adverse events (NCI CTCAE) version 4.03 will be used for all grading. In this study, a DLT will occur if CTCAE grade 4 neutropenia lasts more than 4 consecutive days, if CTCAE grade 3 thrombocytopenia is associated with clinically significant bleeding or if there is grade 4 thrombocytopenia.
Time Frame: Up to 12 months
Population: All participants
Measure: Number; unit: dose in mg
Arm/Group | Tamoxifen and Ribociclib With Goserelin
Number analyzed (Participants) | 7
dose in mg | 400

2. Secondary Outcome: Progression-free Survival (PFS) at Six Months
Description: Occurrence of Progression Survival at 6 months. PFS: On study date to date of progression or the same as overall survival time if not progressed. Progressive Disease (PD): At least a 20% increase in the sum of the longest diameter (LD) of target lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: 6 months
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tamoxifen and Ribociclib With Goserelin
Number analyzed (Participants) | 7
percentage of participants | 57.1 [17.2 to 83.7]

3. Secondary Outcome: Overall Survival (OS) at Six Months
Description: Occurrence of Overall Survival at 6 months. OS: On study date to expired date or last visit date if not deceased.
Time Frame: 6 months
Population: All participants.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tamoxifen and Ribociclib With Goserelin
Number analyzed (Participants) | 7
percentage of participants | 83.3 [27.3 to 97.5]

ADVERSE EVENTS:
Time Frame: 1 year, 2 months
Groups:
- Tamoxifen and Ribociclib With Goserelin: All participants were enrolled and treated on Cohort 1 (Ribociclib 400 mg PO D1-21; Tamoxifen 20 mg PO QD (1) only.
Arm/Group | Tamoxifen and Ribociclib With Goserelin
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 2/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen and Ribociclib With Goserelin (N=7)
Gastrointestinal - Other, Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (3)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tamoxifen and Ribociclib With Goserelin (N=7)
Neutrophil count decreased (Investigations) | 4 (9)
White blood cell decreased (Investigations) | 4 (8)
Alanine aminotransferase increased (Investigations) | 3 (9)
Aspartate aminotransferase increased (Investigations) | 3 (9)
Platelet count decreased (Investigations) | 3 (3)
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 (5)
Alkaline phosphatase increased (Investigations) | 1 (1)
Cholesterol high (Investigations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Weight loss (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (4)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 1 (2)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3)
Dizziness (Nervous system disorders) | 2 (2)
Dysgeusia (Nervous system disorders) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Non-cardiac chest pain (General disorders) | 1 (1)
Otitis media (Infections and infestations) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Cardiac disorders - Other, T Wave Inversion, Q Wave in II, on EKG (Cardiac disorders) | 1 (1)
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Eyelid function disorder (Eye disorders) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (4)
Lymphedema (Vascular disorders) | 1 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-14): https://cdn.clinicaltrials.gov/large-docs/75/NCT02586675/Prot_SAP_000.pdf